CLINICAL TRIAL: NCT04846816
Title: An Open Label, Single Dose Study to Assess Safety and Efficacy of a Novel Patch Infusor Device and Novel SUBCUTaneous Furosemide Formulation Combination in Patients With Heart Failure: a Phase I Clinical Trial
Brief Title: A Study to Assess Safety and Efficacy of a Novel Patch Infusor Device and Novel SUBCUTaneous Furosemide Formulation Combination in Patients With Heart Failure
Acronym: SUBCUT-HF I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SQ Innovation, Inc. (Industry)
Collaborators: University of Glasgow (Other); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN18CA193
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The drug and device combination is called SQIN-01. SQIN-01 is a combination of SQIN-Infusor and SQIN-Furosemide Investigational pump (SQIN-Infusor, medical device) intended for subcutaneous infusion of investigational product, SQINFurosemide.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SQIN-01 (Experimental): The drug and device combination is called SQIN-01. SQIN-01 is a combination of SQIN-Infusor and SQIN-Furosemide Investigational pump (SQIN-Infusor, medical device) intended for subcutaneous infusion of investigational product, SQINFurosemide.
  Interventions: Combination Product: SQIN-01

INTERVENTIONS:
Combination Product: SQIN-01 — The drug and device combination is called SQIN-01. SQIN-01 is a combination of SQIN-Infusor and SQIN-Furosemide Investigational pump (SQIN-Infusor, medical device) intended for subcutaneous infusion of investigational product, SQINFurosemide.

SUMMARY:
This is a single-centre, prospective, open-label, non-comparative clinical trial assessing the on-body performance of an investigational drug delivery device (SQIN-Infusor) in patients hospitalised due to HF.

DETAILED DESCRIPTION:
The investigational product consists of a novel higher concentration (30mg/mL) furosemide formulation developed for subcutaneous administration and a novel patch pump placed on the abdominal skin. This trial will investigate the on body performance of novel patch pump delivering the novel formulation. Study parameters include pharmacokinetic measurements and diuretic response following subcutaneous administration of 80mg of furosemide solution in 2.7mL in patients with heart failure (HF). Recruitment will be restricted to 1 site with a recruitment target of 20 patients. All trial related activities will be conducted in an inpatient environment.

ELIGIBILITY:
Inclusion Criteria:

* • Written informed consent

  * Male or female ≥18 years of age
  * Meet ESC criteria for diagnosis of HF(4)
  * Inpatient with a primary diagnosis of HF requiring treatment with intravenous furosemide at dose

Exclusion Criteria:

* • Unable to consent to inclusion in study due to lack of capacity

  * Requiring treatment with intravenous furosemide at dose >200 mg per day as determined by the usual care team
  * Current inotropes, vasopressors or intra-aortic balloon pump therapy
  * Concomitant use of diuretics in 12 hours preceding administration of study drug with SQIN-Infusor
  * Systolic blood pressure (SBP) <90 mmHg
  * Pregnancy or breastfeeding
  * Left sided valve disease with planned surgery or percutaneous intervention
  * Type 1 myocardial infarction during index hospitalisation (type 2 myocardial infarctions are allowed)(5)
  * Any surgical or medical condition which prevents patient from ambulation during the infusion
  * Renal impairment, defined as eGFR < 30 mL/min/1.73 m2 at screening.
  * Patient on active cardiac transplant waiting list
  * Potassium <3.0 mmol/L
  * Potassium >6.0 mmol/L
  * Sodium <125 mmol/L
  * Any contraindications for furosemide administration as per furosemide SmPC
  * Any surgical or medical conditions, which in the opinion of the investigator may pose an undue risk to the subject, interfere with participation in the study or which may affect the integrity of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
To investigate the safety, tolerability, efficacy and on-body performance of a novel patch infusor device and novel furosemide formulation combination (SQIN-01). | 24 hours from start of infusion
  Safety as determined by treatment emergent adverse events and adverse drug events
Infusion site pain | During 5 hour infusion
  Measured on a scale of 0 = no pain to 10 = most pain
Any device failures | During 5 hour infusion
  Any device failures
Serum furosemide concentration | At baseline
  Serum furosemide concentration
Serum furosemide concentration | At 60 minutes
  Serum furosemide concentration
Serum furosemide concentration | At 240 minutes
  Serum furosemide concentration

SECONDARY OUTCOMES:
Urine volume | 8 hours
  Urine volume (ml) in urine collected 8 hours after start of SQIN-Furosemide infusion
Sodium concentration in urine | 8 hours
  Sodium concentration (mmol) in urine collected 8 hours after start of SQIN-Furosemide infusion
Presence of local skin reactions | After 5 hour infusion
  Presence of local skin reactions on examination
Patient acceptability | After 5 hour infusion
  Patient acceptability using System Usability Scale - from 0 to 100 with a lower number correlating to poor usability and a higher number correlating to better usability by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Petrie, MBChB, Study Chair — University of Glasgow
Locations (1):
- Queen Elizabeth University Hospital, NHS Greater Glasgow & Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
to publish